CLINICAL TRIAL: NCT01807507
Title: Clinical Verification Evaluation of VeinViewer® Device
Status: Completed | Type: Observational
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP1016
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Vein Width
Keywords: Veins; Vascular Access

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Device: VeinViewer

INTERVENTIONS:
Device: VeinViewer — VeinViewer® is designed to improve vascular access treatment standards and provide the highest possible quality in volunteer care. The device is a non-invasive handheld electronic visual aid device designed to project an image of superficial, subcutaneous vascular structures on the surface of the skin. VeinViewer's primary purpose is to assist in vascular visualization for IV starts and blood draws.

SUMMARY:
Measure accuracy of vein width using VeinViewer®, compared against ultrasound imaging as a gold standard

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be able to read and understand English to understand the consent letter

Exclusion Criteria:

* Less than 18 years of age
* Unable to read and understand English to understand the consent letter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Device validation versus ultrasound | Immediately after assessment-Day 1
  The focus of this study is to understand the clinical effectiveness of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Wagner, MS, Principal Investigator — Christie Medical Holdings, Inc.
Locations (1):
- Christie Medical Holdings, Inc., Kitchener, Ontario, Canada